CLINICAL TRIAL: NCT02173574
Title: An Open-label, Two Part Investigation of the Pharmacokinetics, Safety, and Tolerability of Alisporivir and EDP239 When Co-administered to Healthy Adult Subjects
Brief Title: Two-way Interaction Between Alisporivir and EDP239
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDEB025A2119; 2013-004287-59 (EudraCT Number)
Record Dates: First submitted 2014-06-20; First posted 2014-06-25 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Hepatitis C Virus
Keywords: Hepatitis C Virus, Viral, Antiviral, Infection, Infectious disease, alisporivir, EDP239, DEB025
MeSH Terms: conditions — Hepatitis C; Infections; Communicable Diseases | interventions — EDP-239

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-Label Single Arm Cohort (Experimental)
  Interventions: Drug: DEB025; Drug: EDP239

INTERVENTIONS:
Drug: DEB025
Drug: EDP239

SUMMARY:
The purpose of Part 1 is to inform dose selection for use of alisporivir and EDP239 in combination and obtain initial safety data for co-administration of alisporivir and EDP239 to support future treatment studies in patients. The purpose of Part 2 is to inform the drug-drug interaction potential of EDP239 more broadly and possibly facilitate the interpretation of lower than expected alisporivir concentrations in Part 1, if observed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 to 55 years of age
* Body weight at least 50 kg

Exclusion Criteria:

* Women of child bearing potential
* Tobacco use
* History or evidence of any inherited bilirubin disease or disorder, including not not necessarily limited to Dubin-Johnson Syndrome, Gilbert's syndrome, and Rotor Syndrome

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve (AUC) | EDP239 P1: D7/15/21: 0 (pre), and postdose 1,2,3,4,5,6,8,12hr P2: at D10 pre and postdose at 1,2,3,4,5,6,8,12hr,D11/12/13/14. DEB025 P1: D15/21 at pre and postdose at 1,2,3,4,5,6,8,12hr P2: D3/10(Per2) at pre, 0.5,1,2,4,6,8,12,24,3,48,72,96,120,144,168
  The following PK parameters were determined from the plasma concentration time profile of EDP239 and DEB025 using a non-compartmental method: AUCtau: Area under the plasma concentration-time curve from time zero to the end of the dosing interval AUC0-24: Area under the plasma concentration-time curve from time zero to 24 hours AUClast: Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration. AUClast was calculated as the sum of linear trapezoids using non-compartmental analysis. AUCinf: Area under the plasma concentration-time curve from time zero to infinity. AUCinf was calculated by adding AUClast and the value obtained from dividing the last measurable plasma concentration by λz, where λz was determined from automated linear regression of the last three time points with non-zero concentrations in the terminal phase of the log-transformed concentration-time profile
Adverse Events | Part 1: Screening (Day -22 to -2) to Day 35 Part 2: Period 1- Screening (Day -22 to -2) to Day 8 Period 2- Day -1 to 28
  AEs are reviewed on an ongoing basis
Safety Labs | Part 1: Screening (Day -22 to -2), -1, 1, 7, 14, 21 Part 2: Period 1- Screening (Day -22 to -2), Day -1, 8 Period 2- Day -1, 1, 14, 28
  Laboratory samples will be assessed for the following: hematology, blood chemistry, and urinalysis
Plasma Pharmacokinetics (PK) of DEB025 and EDP239: Observed Maximum Plasma Concentration Following Drug Administration at Steady State (Cmax, ss) | EDP239 P1: D7/15/21: 0 (pre), and postdose 1,2,3,4,5,6,8,12hr P2: at D10 pre and postdose at 1,2,3,4,5,6,8,12hr,D11/12/13/14. DEB025 P1: D15/21 at pre and postdose at 1,2,3,4,5,6,8,12hr P2: D3/10(Per2) at pre, 0.5,1,2,4,6,8,12,24,3,48,72,96,120,144,168
  Cmax,ss was directly determined from the raw plasma concentration-time data.
Vital Signs | Part 1: Screening (Day -22 to -2) to Day 35 Part 2: Period 1- Screening (Day -22 to -2) to Day 8 Period 2- Day -1 to 28
  Blood pressure and pulse rate will be assessed for safety.

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- Investigative Site, Berlin, Germany